CLINICAL TRIAL: NCT00632190
Title: Measurement of Fluorescence EEM of Cervical Intraepithelial Neoplasia
Brief Title: Spectroscopy in Diagnosing Dysplasia and Neoplasia in the Cervix in Women Undergoing Colposcopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000581311; BCCR-C99-0441; C99-0441
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Fluorophotometry; Colposcopy

INTERVENTIONS:
Other: fluorophotometry
Procedure: colposcopic biopsy
Procedure: colposcopy
Procedure: light-scattering spectroscopy

SUMMARY:
RATIONALE: New diagnostic procedures, such as spectroscopy, may be a less invasive way to check for dysplasia and neoplasia in the cervix. Spectroscopy may also used as a screening test to help doctors find cervical cancer sooner, when it may be easier to treat.

PURPOSE: This clinical trial is studying how well spectroscopy works in diagnosing dysplasia and neoplasia in the cervix in women undergoing colposcopy or Pap testing.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify potential improvements for a noninvasive method of diagnosing dysplasia and neoplasia in the cervix using fluorescence and reflectance spectroscopy.
* To measure the reflection and fluorescence spectra in vivo of sites in the human cervix.
* To further refine fluorescence spectroscopy for detection of cervical lesions via better classification of normal columnar tissue and non-neoplastic tissue with inflammation, and low- and high-grade squamous intraepithelial lesions.
* Evaluate and validate the wavelength selections for the spectroscopy device derived from in vitro measurements.
* Determine the sensitivity and specificity of this device for the diagnosis of cervical intraepithelial neoplasia.

OUTLINE: This is a multicenter study. Patients are stratified according to menopausal status and current treatment (premenopausal not on oral contraceptive pills [OCP] vs premenopausal on OCP vs postmenopausal not on hormone replacement therapy [HRT] vs postmenopausal on HRT).

* Diagnostic study: As part of routine colposcopic evaluation, patients undergo placement of the probe on 1 to 4 sites in the cervix for 2-5 minutes. Up to two colposcopically abnormal sites and two normal sites are biopsied. Blood is drawn for hormone levels. Fluorescence excitation and emission matrix (EEM) data and reflectance spectroscopic information is acquired from patients with an abnormal Papanicolaou smear.
* Screening study: Fluorescence EEM and reflectance spectroscopic information is acquired from patients with a history of normal Papanicolaou smears.

PROJECTED ACCRUAL: A total of 800 patients with abnormal Papanicolaou smears and 1000 subjects with normal Papanicolaou smears are accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Referred to the Colposcopy clinic at Vancouver General Hospital, the MD Anderson Cancer Center, or the University of Texas at Austin
* Abnormal or normal Papanicolaou smear
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Pre or post-menopausal
* Not pregnant

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Measurement of reflection and fluorescence spectra in vivo of sites in the human cervix
Refinement of fluorescence spectroscopy for detection of cervical lesions via better classification of normal columnar tissue and non-neoplastic tissue with inflammation, and low- and high-grade squamous intraepithelial lesions
Validation of wavelength selections for the spectroscopy device derived from in vitro measurements
Sensitivity and specificity of this device for the diagnosis of cervical intraepithelial neoplasia

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lam — British Columbia Cancer Agency